CLINICAL TRIAL: NCT04194034
Title: A Dose-escalation and Phase IIa Study of TG6002 Plus Flucytosine in Patients With Unresectable Colorectal Cancer With Liver Metastases
Brief Title: Study of Intrahepatic Arterial Infusion of TG6002 in Combination With 5-FC in Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study has been terminated after Phase I part on 23 February 2023
Sponsor: Transgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG6002.03
Record Dates: First submitted 2019-12-08; First posted 2019-12-11 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Flucytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TG6002 and flucytosine (5-FC) combination (Experimental)
  Interventions: Biological: TG6002; Drug: Flucytosine (5-FC)

INTERVENTIONS:
Biological: TG6002 — Phase I part: Dose escalation from 1 x 10E6 PFU to 1 x 10E9 PFU. Phase II part: Established recommended Phase II dose (RP2D).
  Intrahepatic arterial (IHA) administration on Day 1 within a 14-day cycle of TG6002/5-FC combination treatment.
  A second cycle of TG6002/5-FC combination starting with TG6002 (IHA) administration at the same dose on Day43 can be initiated if no progressive disease or Dose Limiting Toxicity event in between; maximum 2 cycles of TG6002/5-FC combination treatment for each patient.
Drug: Flucytosine (5-FC) — Oral administration 4 times per day at the total dose of 200 mg/kg/day for 10 consecutive days per 14-day cycle of TG6002/5-FC combination.
  A second cycle of TG6002/5-FC combination will be initiated if no progressive disease or Dose Limiting Toxicity event in between.

SUMMARY:
This study will include two parts:

* Phase I part is a dose-escalation study to assess the safety of increasing doses of TG6002 in combination with oral flucytosine (5-FC) in consecutive cohorts of 3 to 6 patients with colorectal cancer and unresectable liver metastases according to a 3+3 design
* Phase IIa part is an extension of the phase I part at the recommended phase II dose to evaluate the efficacy of TG6002 in combination with oral flucytosine (5-FC) in patients with colorectal cancer and unresectable liver metastases.

In both parts, tumor response will be evaluated on local assessment using RECIST 1.1.

All patients will be followed until disease progression, death due to any cause or the date of data cut-off, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable metastatic CRC with at least one measurable liver metastasis
2. At least one liver metastasis amenable to biopsy
3. Patients previously exposed to fluoropyrimidine-based chemotherapy
4. (Phase I) Patients having failed, are intolerant to, or unsuitable for both oxaliplatin and irinotecan-based chemotherapy, or, in the UK only, patients on or entering a period of clinical observation without treatment
5. (Phase IIa) Patients having failed, are intolerant to, or unsuitable for both oxaliplatin and irinotecan-based chemotherapy.
6. Aged ≥18 years
7. Estimated life expectancy >3 months
8. ECOG performance status ≤1

Exclusion Criteria:

1. Predominant extrahepatic disease
2. Symptomatic brain metastases or meningeal tumors
3. Any contraindication to intrahepatic artery infusion procedure
4. Received other investigational therapy or had surgery within 4 weeks of treatment initiation which would interfere with study treatment
5. Received locoregional therapy for CRC within 4 weeks prior to treatment initiation
6. Severe uncontrolled coagulopathy OR anticoagulant medication
7. Antiviral therapy active on vaccinia virus, e.g., ribavirin, interferon/pegylated interferon
8. Immunosuppression due to immunosuppressive medication including steroids equivalent to prednisolone >10mg/day taken for more than 4 weeks within 3 months prior to TG6002 treatment initiation
9. Patients treated with 3 or more anti-hypertensive agents AND/OR patients with signs of advanced hypertensive disease, such as left ventricular hypertrophy, hypertensive encephalitis or history of hemorrhagic stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (Phase I part) | Day 28
  Incidence of Adverse events using CTCAE v5.0
Disease Control Rate (Phase II part) | Week 10
  Proportion of patients whose tumour assessment is either complete response (CR), partial response (PR), or stable disease (SD)

CONTACTS AND LOCATIONS:
Locations (3):
- France (2):
  - Centre Léon Bérard, Lyon
  - Institut Gustave Roussy, Villejuif
- NHS St James's University Hospital, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No